CLINICAL TRIAL: NCT07356544
Title: HER2 in Advanced NSCLC: an Observational, Prospective, Multi-centric Study Exploring HER2 Mutations Incidence and Therapeutic Management in Italy. The HEROS Study - GOIRC-01-2022
Brief Title: Observational, Prospective, Multi-centric Study Exploring HER2 Mutations Incidence and Therapeutic Management in aNSCLC
Acronym: HEROS
Status: Recruiting | Type: Observational
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: GOIRC-01-2022
Record Dates: First submitted 2025-01-14; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-01

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); HER2
Keywords: HER2 mutated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE material and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The HEROS study is an Italian observational multicenter prospective study aimed to investigate the current diagnostic and therapeutical approach towards HER2 mutated NSCLC in clinical practice. The enrolment will start in September 2024 until September 2025. A 12-months follow-up window will be performed.

DETAILED DESCRIPTION:
The HEROS study will be conducted in partnership with ATLAS project: all patients prospectively enrolled in ATLAS project will be used to fulfil primary and secondary objectives. Information will be obtained by querying ATLAS database (59 centers) in aggregated manner. ATLAS project is a multi-centric retrospective/prospective Italian study aimed to describe prevalence of different oncogene alterations in all new diagnosed advanced NSCLC patients (5,000 patients/year). In particular, prevalence of HER2-mutated patients will be calculated on all patients enrolled in ATLAS project. Approximately 100 HER2 mutated patients enrolled in ATLAS study will be studied for secondary and explorative objectives. Moreover, a subset of centers (25 centers) will enrol patients also for Prospective Biomarker Analysis in order to perform exploratory analysis on blood and tissue samples according to the availability of tissue specimens from the primary tumor or metastatic sites. All centers that will participate for Prospective Biomarker Analysis necessarily will be included into ATLAS project.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 (Prevalence study population)

1. Male or female, aged at least 18 years.
2. Pathologically confirmed diagnosis of NSCLC from September 2024 to September 2025.
3. Locally advanced (IIIC), not amenable to multimodal approach (chemo-radiotherapy), or metastatic (IV) NSCLC according to TNM VIII edition.
4. Enrolled in ATLAS project. Cohort 2 (HER2 mutations study population)
5. Included in Cohort 1.
6. Presence of HER2 mutation.
7. Enrolled in ATLAS project. Cohort 3 (Prospective Biomarker Analysis population)
8. Included in Cohort 2.
9. Availability of tissue sample from the first 50 patients enrolled in cohort 2.
10. Written informed consent (HEROS project) must be obtained before any study-related procedure.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-mutated advanced non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HER2 mutation | 1 year
  Percentage of advanced NSCLC with HER2 mutations in Italy clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Tiseo, MD, PhD, Study Director — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (22):
- Italy (22):
  - IRCCS "Giovanni Paolo II", Bari, BA
  - Istituto Romagnolo per lo Studio dei Tumori IRST "Dino Amadori", Meldola, FC
  - Arcispedale Sant'Anna, Ferrara, FE
  - Ospedale Policlinico San Martino, Genova, GE
  - Ospedale Versilia, Lido di Camaiore, LU
  - Azienda Sanitaria Toscana Nord - Ovest, Lucca, LU
  - IRCCS San Gerardo dei Tintori, Monza, MB
  - IRCCS Ospedale San Raffaele, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Istituto Clinico Humanitas IRRCS, Rozzano, MI
  - Azienda Ospedaliero - Universitaria di Modena, Modena, MO
  - Istituto Oncologico Veneto IRCCS, Padua, PD
  - Azienda Ospedaliera di Perugia, Perugia, PG
  - Centro di Riferimento Oncologico IRCCS di Aviano, Aviano, PN
  - Azienda Ospedaliera - Universitaria di Parma, Parma, PR
  - Fondazione IRCCS Policlinico S. Matteo, Pavia, PV
  - Azienda Ospedaliero - Universitaria di Reggio Emilia, Reggio Emilia, RE
  - Istituto Nazionale dei Tumori Regina Elena IRCCS - IFO, Roma, RM
  - Azienda Ospedaliera San Camillo Forlanini, Roma, RM
  - AOU San Luigi Orbassano, Orbassano, TO
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC), Udine, UD
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona, VR

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT07356544/Prot_SAP_000.pdf